CLINICAL TRIAL: NCT05144334
Title: An Open Label, Escalating Multiple Dose Study to Evaluate the Safety, Toxicity, Pharmacokinetics, and Preliminary Activity of BTX-1188 in Subjects With Advanced Malignancies
Brief Title: A Study of BTX-1188 in Subjects With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Biotheryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTX-1188-001
Record Dates: First submitted 2021-11-09; First posted 2021-12-03 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor; Non Hodgkin Lymphoma; Acute Myeloid Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- BTX-1188 Dose Cohort 1 (Experimental): Starting dose of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188
- BTX-1188 Dose Cohort 2 (Experimental): First dose escalation of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188
- BTX-1188 Dose Cohort 3 (Experimental): Second dose escalation of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188
- BTX-1188 Dose Cohort 4 (Experimental): Third dose escalation of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188
- BTX-1188 Dose Cohort 5 (Experimental): Fourth dose escalation of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188
- BTX-1188 Dose Cohort 6 (Experimental): Fifth dose escalation of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188
- BTX-1188 Dose Cohort 7 (Experimental): Sixth dose escalation of BTX-1188 administered orally per dosing schedule
  Interventions: Drug: BTX-1188

INTERVENTIONS:
Drug: BTX-1188 — One 28 day cycle of treatment will consist of 4 weeks of treatment with BTX-1188 administered orally per dosing schedule.

SUMMARY:
This is a multicenter, open label, nonrandomized, sequential dose escalation, multiple dose study designed to evaluate the safety, toxicity, and pharmacokinetics (PK) as well as preliminary efficacy of BTX-1188 orally administered in subjects with advanced malignancies.

DETAILED DESCRIPTION:
Study BTX-1188-001 is a multicenter, open label, nonrandomized, sequential dose escalation study to evaluate the safety, toxicity, PK, and preliminary efficacy of BTX-1188. Dose escalation will be conducted in subjects with acute myeloid leukemia (AML) and advanced lymphoid and solid tumors. Based on the results of the dose escalation, a recommended Phase 2 dose will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Demonstration of understanding and voluntarily signing of an informed consent form
* Age ≥ 18 years
* Part A - Relapsed or refractory AML, according to the World Health Organization (WHO) classification (Arber, Orazi, et al., 2016). Subjects must be ineligible for or have exhausted standard therapeutic options that would otherwise be likely to provide clinical benefit. Part B - B cell NHL that is refractory to or intolerant of all standard therapy or for which no standard therapy is available or histologically or cytologically documented, incurable or metastatic solid tumor that has failed all available standard therapies with known benefit.
* Subjects with solid tumors must have measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). NHL subjects must have bi-dimensionally measurable disease on cross sectional imaging by computed tomography (CT) or magnetic resonance imaging (MRI) as defined by Lugano criteria (Cheson, Fisher, et al., 2014).
* Adequate organ function
* Females must avoid pregnancy for at least 4 weeks before beginning BTX-1188 therapy, during therapy, during dose interruptions, and for at least 4 weeks after completing therapy and agree to either abstain from sexual intercourse or use two highly effective methods of contraception (for up to 4 weeks after last dose of study drug)
* Males sexually active with a woman of childbearing age must agree to use barrier method of birth control during and after the study and not donate sperm (for up to 4 weeks after last dose of study drug).

Exclusion Criteria:

* Life expectancy <3 months, as determined by the Investigator.
* Treatment with any local or systemic antineoplastic therapy (including chemotherapy, hormonal therapy, or radiation) within 3 weeks prior to first dose of BTX-1188
* Immediate life-threatening severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Major trauma or major surgery within 4 weeks prior to first dose of BTX-1188.
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤1 except for alopecia or Grade ≤2 immunotherapy-related thyroid toxicity.
* History of, or known, central nervous system (CNS) disease involvement, or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity.
* Clinically significant cardiac disease
* Active uncontrolled systemic fungal, bacterial, mycobacterial, or viral infection
* Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)
* Active hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Second primary malignancy that has not been in remission for greater than 3 years
* Any serious underlying medical (e.g., pulmonary, renal, hepatic, gastrointestinal, or neurological) or psychiatric condition (e.g., alcohol or drug abuse, dementia or altered mental status) or any issue that would limit compliance with study requirements
* Pregnant, lactating, or breastfeeding.
* Participation or plans to participate in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] with BTX-1188 in subjects with advanced malignancies | From first dose of BTX-1188 through 30 days after the last BTX-1188 treatment
  To examine the incidence of clinical and laboratory adverse events after multiple doses of BTX-1188
To determine the recommended Phase 2 dose (RP2D) of BTX-1188 in subjects with advanced malignancies | At the end of Cycle 1 (each cycle is 28 days)
  To assess number of patients experiencing dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Maximum Plasma Concentration of BTX-1188 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, and 8 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the maximum observed concentration (Cmax) after single and repeated oral, once daily doses of BTX-1188
Peak Plasma Concentration of BTX-1188 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, and 8 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the observed time of peak concentration (Tmax) after single and repeated oral, once daily doses of BTX-1188
Area under the plasma concentration of BTX-1188 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, and 8 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the area under the curve (AUC) plasma-concentration after single and repeated oral, once daily doses of BTX-1188.
Half-life of BTX-1188 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, and 8 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the half-life of BTX-1188 after single and repeated oral, once daily doses of BTX-1188.
Objective response rate (ORR) | Up to 2 years after the last treatment or upon death.
  To evaluate the objective response rate (ORR) as determined by the specific disease response criteria.
Best response | For subjects with AML, response will be evaluated at the end of each cycle (each cycle is 28 days) and after the last dose of BTX-1188 (approximately 36 months). For subjects with NHL or solid tumors, response will be evaluated every 8-weeks.
  To evaluate the complete remission/response [CR], CR with incomplete blood count recovery [CRi], morphologic leukemia free state [MLFS], partial remission/response [PR], stable disease or progression as determined by the specific disease response criteria.
Disease Control Rate (DCR) | For subjects with AML, response will be evaluated at the end of each cycle (each cycle is 28 days) and after the last dose of BTX-1188 (approximate 36 months). For subjects with NHL or solid tumors, response will be evaluated every 8-weeks.
  To evaluate the DCR (response + stable disease) as determined by the specific disease response criteria.
Duration of response (DoR) | Up to 2 years after the last treatment or upon death.
  To evaluate the duration of response (DoR), defined as time from the date of first documentation of response to the date of the first documentation of progressive disease (PD), or death due to any cause.
Progression free survival (PFS) | Up to 2 years after the last treatment or upon death.
  To examine the the progression free survival (PFS), defined as time from the date of first dose of study treatment to the first date of documentation of PD, or death due to any cause.
Overall survival (OS) | Up to 2 years after the last treatment or upon death.
  To examine the overall survival (OS), defined as time from the date of first dose of study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Lawhon, Study Director — Biotheryx, Inc.
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas